CLINICAL TRIAL: NCT06696807
Title: The Effects of Immunomodulatory Therapy in Patients with Vasospastic Angina
Brief Title: Immunomodulatory Therapy & VSA
Status: Completed | Type: Observational
Sponsor: Dao Wen Wang (Other)
Responsible Party: Sponsor-Investigator, Dao Wen Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20211259
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Vasospastic Angina
Keywords: Immunomodulatory therapy; vasospastic angina; Cohort Study
MeSH Terms: conditions — Angina Pectoris, Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- traditional therapy group: who received nitrate esters, CCBs, anti-platelet agents, and statins
- immunomodulatory therapy group: who received glucocorticosteroids and/or IVIG in addition to traditional therapy.
  Interventions: Drug: glucocorticosteroids and/or intravenous immunoglobulin

INTERVENTIONS:
Drug: glucocorticosteroids and/or intravenous immunoglobulin — methylprednisolone: 20-200mg/day intravenous immunoglobulin: 5-20 g/day
  Groups: immunomodulatory therapy group

SUMMARY:
Vasospastic angina (VSA) is caused by brief spasms of the main coronary artery and its major branches, resulting in varying degrees of luminal occlusion. Although vasodilator therapy is widely used and significantly alleviates VSA symptoms, it has not led to notable improvements in the prognosis of patients with VSA. Recent studies have suggested that inflammation plays a crucial role in VSA. This study aimed to evaluate the potential effectiveness of immunomodulatory therapy for improving patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

(1) Transient total or subtotal occlusion of the coronary artery (contraction >90%) observed either spontaneously or in response to irritant stimulation (typically acetylcholine, ergot, or hyperventilation); (2) Presence or absence of ischemic electrocardiogram changes during episodes; (3) Nitrate-responsive angina during spontaneous episode: rest angina and/or marked diurnal variation in exercise tolerance and/or episodes precipitated by hyperventilation and/or suppression of episodes by calcium channel blockers.

Exclusion Criteria:

(1) age 15 years or older; and (2) suspected VSA with chest pain and evidence of coronary spasm, or VSA diagnosed intraoperatively or at discharge.

The following exclusion criteria were applied: (1) failure to meet the diagnostic criteria for VSA; (2) presence of aortic disease, cardiomyopathy, malignant tumor, Kounis syndrome, or other diseases that may affect the outcome; (3) insufficient clinical data available; and (4) loss to follow-up.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 160 participants with suspected VSA between October 2018 and April 2024 were selected. After the screening process, 71 participants were included in the analysis. The participants were divided into two groups according to the treatment received, with 50 and 21 participants in the traditional and immunomodulatory therapy groups, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
adverse outcomes | From Feb 2017 to Feb 2024
  readmissions due to the onset of coronary spasm or VSA, MACE (including non-fatal stroke, non-fatal myocardial infarction, cardiovascular death) and all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
We are working hard to have IPD sharing plan and are willing to share it with other researchers.